CLINICAL TRIAL: NCT05067803
Title: Pilot Study for the Assessment of the Quality of Echocardiography Exam When Obtained by Novice Users While Using the USEG Software.
Brief Title: Study for the Assessment of USEG Software.
Status: Completed | Type: Observational
Sponsor: UltraSight (Industry)
Responsible Party: Sponsor
Other Study IDs: USEG-101
Record Dates: First submitted 2021-09-23; First posted 2021-10-05 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-02

CONDITIONS: Cardiac Disease
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The product is comprised of software that aids in automated guided ultrasound image acquisition for novice users (medical professional without experience in performing echocardiography, e.g. nurses, physicians assistants, medical doctors, medical student etc.).

The software provides real-time feedback during image acquisition to optimize image capture and determine whether image quality is sufficient for medical evaluation. The software is designed to be used with any echocardiographic ultrasound system. The Philips Lumify hand-held ultrasound device will be used for this study.

* Images can be acquired manually by a novice user.
* Each novice user will have a training course of 8 hours, before the study commences.

DETAILED DESCRIPTION:
Study Design:

This pilot study is a single center, multi-reader multi-case study, primarily designed to obtain the quality of the echocardiography exam, obtained by novice users when using the USEG software.

Eligible subject will undergo the examination twice on a single study visit : once by one of novice users when using the USEG software and once by one of the expert sonographers without the aid of the software.

Each novice user will perform the examination on approximately 30 subjects (depending on the number of novice user, with the aim that the number of examinations by each novice will be the same).

The assignment of the novice user and expert sonographer to subjects and their order within a subject will be based upon their availability once the subject's is enrolled. In case of more than 1 available novice, the exam will be assigned to the novice with the least exams performed so far.

At least 10 subjects will be enrolled from each of the following three BMI groups= < 25; =25 to <30; => 30.

Study Procedures:

After an informed consent is obtained, screening was completed and eligibility has been confirmed, each subject will undergo the examination twice on the day of visit (Day 1): once by a novice user and once by an expert sonographer.

In case of any administrative delay, the investigator may address the issue with the sponsor, and upon approval, the second examination may be postponed in up to 96 hours.

The novice user will obtain at least 10 clips using the UltraSight guidance software for 10 pre-defined views from each patient, and an expert sonographer will obtain 10 clips for the same at least 10 views without the aid of the UltraSight software.

The order in which the novice user and expert sonographer performs the examination per patient will be based on their availability once the subject's is enrolled. In case of more than 1 available novice, the exam will be assigned to the novice with the least exams performed so far.

Adverse events will be monitored throughout the visit.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and older
2. Subjects willing and able to give written informed consent.

Exclusion Criteria:

1. Emergency (non-elective) admission within 24 h prior to participating in the study
2. Female subjects who are pregnant (WOCBP* will perform a urine pregnancy test)
3. Unable to lie as required in all the classic positions for standard TTE exam: supine on back / left decubitus.
4. Subjects who currently participate a clinical trial, involving interventional cardiac devices
5. Subjects who have prior Echo exam with description of Low/Poor quality exam in the echo report
6. Subjects with BMI above 40
7. Subjects experiencing a known or suspected acute cardiac event
8. Subjects with severe chest wall deformity as per previous medical records and physical examination
9. Subjects who have undergone pneumonectomy
10. Subjects whose anatomy does not lend itself to yield diagnosable echocardiography clips (i.e. situs inversus with dextrocardia, single ventricle anatomy due to congenital heart defect, etc.)

    * A woman is of childbearing potential if she is postmenarchal, has not reached a postmenopausal state (≥12 continuous months of amenorrhea with no identified cause other than menopause), and is not permanently infertile due to surgery (i.e., removal of ovaries, fallopian tubes, and/or uterus) or another cause as determined by the investigator (e.g., Müllerian agenesis.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Up to 100 male and female adults confirmed as eligible according to eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2021-12-24 (Actual); Primary Completion 2022-01-23 (Actual); Study Completion 2022-01-23 (Actual)

PRIMARY OUTCOMES:
To assess the quality of clips obtained by novice users when using the USEG software. | 1 year.
  The expert cardiologists will evaluate whether the echo examination has sufficient to evaluate each of the primary endpoints:
  1. Sufficient quality to assess Left Ventricular (LV) size: (YES/NO)
  2. Sufficient quality to assess LV function: (Yes/No)
  3. Sufficient quality to assess Right Ventricular size: (Yes/No)
  4. Sufficient quality to assess presence of non-trivial pericardial effusion: (Yes/No)

SECONDARY OUTCOMES:
Sufficient quality assessment for six (6) anatomic elements. | 1 year.
  The expert cardiologists will evaluate whether the echo examination has sufficient quality to evaluate the following six (6) anatomic elements:
  1. Qualitative visual assessment of RV function: (Yes/No)
  2. Qualitative visual assessment of left atrium size: (Yes/No)
  3. Qualitative visual assessment of Aortic valve structure: (Yes/No)
  4. Qualitative visual assessment of Mitral valve structure: (Yes/No)
  5. Qualitative visual assessment of Tricuspid valve structure: (Yes/No)
  6. Qualitative visual assessment of IVC size: (Yes/No)
Diagnostic quality assessment. | 1 year.
  The expert cardiologists will evaluate if each of the following 10 views can be considered of diagnostic quality:
  * Apical 4 chamber
  * Apical 2 chamber
  * Apical 3 chamber
  * Apical 5 chamber
  * Para Sternal Long Axis
  * Para Sternal short axis - Aortic Valve (AV)
  * Para Sternal short axis - Mitral Valve (MV)
  * Para Sternal short axis - Papillary Muscle (PM)
  * Sub Costal - 4 chamber
  * Sub Costal - Inferior Vena Cava (IVC)f

OTHER OUTCOMES:
Safety outcome. | 1 year.
  Adverse Events.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Klempfner, MD, Principal Investigator — Sheba MC; Danny Spiegelstein, MD, Study Director — UltraSight
Locations (1):
- Sheba MC, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No